CLINICAL TRIAL: NCT02227082
Title: Olaparib Dose Escalation in Combination With High Dose Radiotherapy to the Breast Andregional Lymph Nodes in Patients With Breast Cancer
Brief Title: Olaparib and Radiotherapy in Inoperable Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N13ORB; 2011-001586-40 (EudraCT Number)
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Malignant Neoplasm; Inflammatory Breast Carcinoma; Triple-Negative Invasive Breast Carcinoma
Keywords: radiotherapy; olaparib; breast cancer; locally advanced breast cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms | interventions — Radiotherapy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy and olaparib (Experimental): radiotherapy: 61.18 Gy olaparib: dose escalating
  Interventions: Radiation: radiotherapy; Drug: olaparib

INTERVENTIONS:
Radiation: radiotherapy — The whole breast and regional lymph nodes will receive 23 x 2.03 Gy per fraction (total 46.69 Gy) At the macroscopic tumor a added SIB will be given of 23 x 0.63Gy . Total dose: 61.18 Gy
Drug: olaparib — The pre-defined dose levels of olaparib are 25mg QD, 25, 50, 100, 200, 300 and 400 mg BID
  Other Names: AZD2281; KU-0059436

SUMMARY:
The majority of breast cancer patients receive radiotherapy as part of their treatment. Radiotherapy improves both locoregional control and overall survival. In most patients with breast cancer the locoregional recurrence rate (LRR) is low, however still high LRRs are found in certain patient groups, especially in locally advanced, inflammatory and triple negative breast cancer. Olaparib is a potent PARP inhibitor developed as an anti-cancer drug for homologous recombination (HR) defected tumors and as a dose intensifier for chemo- and radiotherapy. The combination of olaparib and radiotherapy is expected to improve locoregional control and thereby overall survival in both breast cancer patients with a high probability of locoregional recurrence and patients with HR deficient tumors. However, this combination treatment has never been tested in humans before. The purpose of this study is to determine the safety and tolerability of radiotherapy to the breast and regional lymph nodes with concurrent olaparib.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histological proven breast cancer or local recurrence of breast cancer which is inoperable or/and metastatic, including inflammatory breast cancer
* No participation in trial with neoadjuvant systemic treatment, except for previous contralateral breast cancer
* Tumor in breast accessible for biopsy
* WHO performance 0-2
* Life expectancy of at least 6 months
* Adequate hematological, renal and hepatic functions
* Hemoglobin 6.2 mmol/l
* Leucocytes 3.0 x 10E9/l

  * Absolute neutrophil count 1.5x10E9/l
  * Platelet count 100 x 10E9/l
  * Total bilirubin ≤ 1.5 x ULN
  * ASAT/ALAT ≤ 2.5 x ULN; or in the presence of liver metastases ≤ 5 x ULN
  * Creatinine clearance 50 ml/min; measured or calculated
* Evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 21 days of study treatment. Non-childbearing potential or postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * LH and FSH levels in post menopausal range for women under 50 years of age
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilisation (bilateral oophorectomy or hysterectomy)
* Patients of reproductive potential must agree to practice two effective medically approved contraceptive method during the trial and 3 months afterwards
* Signed written informed consent

Exclusion Criteria:

* Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within 3 weeks prior to start of therapy (or a longer period depending on the defined characteristics of the agents used e.g. 6 weeks for mitomycin ornitrosourea). Patient may continue the use of tamoxifen, aromatase inhibitor and LHRH agonists for cancer; bisphosphonates for bone disease and corticosteroids. The use of denosumab for bone disease is not allowed.
* Major surgery within two weeks of starting study treatment.
* Participation in other trial with investigational drug or treatment modality
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required.
* Prior ipsilateral radiotherapy to the chest or breast.
* Blood transfusion in the four weeks prior to study entry
* Persistent toxicities (CTC ≥ grade 2) with the exception of alopecia, caused by previous cancer therapy
* QT-interval > 470 msec
* Significant cardiovascular disease as defined by

  * History of congestive heart failure defined as NYHA class III
  * History of unstable angina pectoris or myocardial infarction up to 3 months prior to trial entry;
  * Presence of severe valvular heart disease
  * Presence of a ventricular arrhythmia requiring treatment;
  * Uncontrolled hypertension
* Patients considered a poor medical risk due to:

  * non-malignant systemic disease
  * active, uncontrolled infection requiring parenteral antibiotics
  * a serious, uncontrolled medical disorder; examples include, but are not limited to:

    * uncontrolled major seizure disorder
    * unstable spinal cord compression
    * superior vena cava syndrome
    * extensive bilateral lung disease on HRCT scan
    * any psychiatric disorder that prohibits obtaining informed consent.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
* Patients with known active hepatic disease (i.e. Hepatitis B or C)
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or features suggestive of MDS/AML on peripheral blood smear.
* Gastrointestinal disorders that may interfere with absorption of the study drug or patients who are not able to take oral medication
* Concomitant medications:

  * Any previous treatment with a PARP inhibitor, including Olaparib
  * Patients receiving the following classes of inhibitors of CYP3A4 (see Section 6.4.2 for guidelines and wash out periods)

    * Azole antifungals
    * Macrolide antibiotics
    * Protease inhibitors
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product
* Breast-feeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicities. | 1 year

SECONDARY OUTCOMES:
Acute toxicity | 3 months after treatment
  severity, duration and relation with treatment of all adverse events according to CTCAE version 4.03 occurring from start of treatment until 3 months after end of treatment
Late toxicity | 3 months until 2 years after end of treatment
  severity, duration and relation with treatment of all adverse events that are possibly, probably or definitely related to the combination treatment according to CTCAE version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Gabe Sonke, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; Marcel verheij, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- [Derived] de Haan R, van Werkhoven E, van den Heuvel MM, Peulen HMU, Sonke GS, Elkhuizen P, van den Brekel MWM, Tesselaar MET, Vens C, Schellens JHM, van Triest B, Verheij M. Study protocols of three parallel phase 1 trials combining radical radiotherapy with the PARP inhibitor olaparib. BMC Cancer. 2019 Sep 10;19(1):901. doi: 10.1186/s12885-019-6121-3. PMID 31500595